CLINICAL TRIAL: NCT00000754
Title: A Randomized Phase II Study of Two Doses of Interferon Alfa-2a (IFN Alfa-2a) in Combination With Zidovudine (AZT) and Dideoxycytidine (ddC) Versus AZT and ddC Only in Patients With HIV Infection and Less Than 400 CD4 Cells/mm3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 197; 11173 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Interferon-alpha
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Interferon alpha-2; Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Interferon alfa-2a
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
To determine the safety and efficacy of two doses of interferon alfa-2a ( IFN alfa-2a ) in combination with zidovudine ( AZT )/zalcitabine ( ddC ) versus AZT/ddC only in patients with HIV infection and CD4 count < 400 cells/mm3.

AZT and ddC inhibit HIV by acting as reverse transcriptase chain terminators, while IFN alfa-2a inhibits translation of viral proteins. Combining agents that act at different sites of viral replication may improve HIV inhibition and produce more effective and sustained anti-HIV effects.

DETAILED DESCRIPTION:
AZT and ddC inhibit HIV by acting as reverse transcriptase chain terminators, while IFN alfa-2a inhibits translation of viral proteins. Combining agents that act at different sites of viral replication may improve HIV inhibition and produce more effective and sustained anti-HIV effects.

Patients are randomly assigned to one of three treatment arms to receive AZT/ddC alone or combined with one of two doses of IFN alfa-2a. Treatment continues for up to 12 months after enrollment of the last patient. Patients are followed at 2, 4, and 8 weeks and every 8 weeks thereafter. Mean duration of follow-up is expected to be 13 months.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Isoniazid for < grade 2 peripheral neuropathy (if patient is also taking 50 mg/day pyridoxine).
* Phenytoin for < grade 2 peripheral neuropathy.
* A 21-day course of adjuvant systemic corticosteroid therapy for moderate to severe Pneumocystis carinii pneumonia (PCP).
* Chemoprophylaxis for PCP, candidiasis, herpes simplex infection (up to 1 g acyclovir daily), and Mycobacterium tuberculosis.

Patients must have:

* HIV infection.
* CD4 count < 400 cells/mm3 within 30 days prior to study entry.

NOTE:

* Minimal Kaposi's sarcoma is allowed.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Active opportunistic infection requiring acute therapy.
* Need for maintenance therapy for cytomegalovirus infection, toxoplasmic encephalitis, or mycobacterial infection.
* Malignancy (other than minimal Kaposi's sarcoma) requiring therapy.
* Grade 2 or worse peripheral neuropathy.

Concurrent Medication:

Excluded:

* Other antiretroviral drugs, biologic response modifiers, cytotoxic chemotherapy, or investigational drugs (unless approved by the protocol chairs).
* Recombinant erythropoietin, G-CSF, or GM-CSF.
* Drugs that cause peripheral neuropathy, e.g., gold, hydralazine, nitrofurantoin, vincristine, cisplatin, disulfiram, and diethyldithiocarbamate (unless approved by the protocol chairs).

Concurrent Treatment:

Excluded:

* Radiation therapy (unless approved by the protocol chairs).

Patients with the following prior conditions are excluded:

* History of intolerance to AZT at 600 mg/day or less.
* Unexplained temperature of 38.5 degrees C persisting for 14 days or longer.
* Unexplained, chronic diarrhea defined as 3 or more stools per day persisting for 14 days or longer.

Prior Medication:

Excluded:

* Acute therapy for opportunistic infection within 14 days prior to study entry.
* Prior ddC, ddI, or IFN alfa-2a.

Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Study Completion 1995-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fischl MA, Study Chair; Richman DD, Study Chair
Locations (4):
- United States (4):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - Ucsd, Avrc Crs, La Jolla, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - Univ. of Miami AIDS CRS, Miami, Florida

REFERENCES:
- [Background] Fischl MA, Richman DD, Saag M, Meng TC, Squires KE, Holden-Wiltse J, Meehan PM. Safety and antiviral activity of combination therapy with zidovudine, zalcitabine, and two doses of interferon-alpha2a in patients with HIV. AIDS Clinical Trials Group Study 197. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Dec 1;16(4):247-53. doi: 10.1097/00042560-199712010-00005. PMID 9402071